CLINICAL TRIAL: NCT06704490
Title: Analysis of the Incidence and Risk Factors of Chronic Pain After Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Professor, Huazhong University of Science and Technology
Other Study IDs: chronic postoperative pain
Record Dates: First submitted 2024-03-18; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain; Cesarean Section Surgery
Keywords: postoperative pain; chronic postoperative pain; cesarean section surgery; Postpartum depression
MeSH Terms: conditions — Pain, Postoperative; Depression, Postpartum | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean section surgery: Observational research
  Interventions: Other: Cesarean section

INTERVENTIONS:
Other: Cesarean section — Observational study without intervention

SUMMARY:
Persistent postoperative pain is a globally recognized issue that deserves attention. Cesarean section is one of the surgeries that may cause persistent postoperative pain. PSPP may affect communication between mother and baby, and may lead to postpartum depression, which has a negative impact on the daily activities and quality of life of mothers. It is an important clinical issue.

The main purpose of this study is to (1) prospectively investigate the overall incidence and characteristics of persistent pain after cesarean section at 3, 6, and 12 months after surgery; (2) Use regression analysis and data modeling analysis to evaluate the relationship between perioperative variables and chronic pain in postpartum women undergoing cesarean section; (3) Analyze the relationship between chronic pain after cesarean section and postpartum depression in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 20 to 50 years old;
* ASA grades I to III;
* Full term pregnancy and planned cesarean section with transverse incision in the lower segment of the uterus;
* Pregnant women who are willing to participate in this study and sign informed consent forms.

Exclusion Criteria:

* Have a history of dementia, mental illness, or any central nervous system disorder;
* Pregnant women who are addicted to alcohol and drugs;
* Difficulty in follow-up or poor patient compliance;
* Has taken other investigational drugs or participated in other clinical trials in the three months prior to being selected for the study;
* Serious complications occur during delivery;
* Unable to cooperate with the research for any reason.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women planning to undergo cesarean section surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain after caesarean section | 2024-01-01-2025-01-01
  Assessment of chronic postoperative pain by Brief Pain Inventory from 0 to ten, The higher the score, the stronger the pain

SECONDARY OUTCOMES:
Identification of high-risk factors for postoperative inadequate analgesia and PONV in obstetric patients based on machine learning methods | 2024-2026
  Postoperative pain is represented by NRS score (0-10). The higher the NRS score, the more severe the pain. A NRS score of ≥ 4 is considered insufficient postoperative analgesia. Analyzed the predictive value of 42 variables, including preoperative, intraoperative, and postoperative variables, for postoperative inadequate analgesia.
Adverse effects of postoperative analgesia | 2024-2026
  Incidence and the risk factors of adverse effects of postoperative analgesia, especially postoperative nausea and vomiting
Checklist for Chronic pain after cesarean section | 2024-2026
  Types of chronic pain after cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Betran AP, Temmerman M, Kingdon C, Mohiddin A, Opiyo N, Torloni MR, Zhang J, Musana O, Wanyonyi SZ, Gulmezoglu AM, Downe S. Interventions to reduce unnecessary caesarean sections in healthy women and babies. Lancet. 2018 Oct 13;392(10155):1358-1368. doi: 10.1016/S0140-6736(18)31927-5. PMID 30322586
- [Result] Klemetti R, Che X, Gao Y, Raven J, Wu Z, Tang S, Hemminki E. Cesarean section delivery among primiparous women in rural China: an emerging epidemic. Am J Obstet Gynecol. 2010 Jan;202(1):65.e1-6. doi: 10.1016/j.ajog.2009.08.032. Epub 2009 Oct 12. PMID 19819416
- [Result] Lumbiganon P, Laopaiboon M, Gulmezoglu AM, Souza JP, Taneepanichskul S, Ruyan P, Attygalle DE, Shrestha N, Mori R, Nguyen DH, Hoang TB, Rathavy T, Chuyun K, Cheang K, Festin M, Udomprasertgul V, Germar MJ, Yanqiu G, Roy M, Carroli G, Ba-Thike K, Filatova E, Villar J; World Health Organization Global Survey on Maternal and Perinatal Health Research Group. Method of delivery and pregnancy outcomes in Asia: the WHO global survey on maternal and perinatal health 2007-08. Lancet. 2010 Feb 6;375(9713):490-9. doi: 10.1016/S0140-6736(09)61870-5. Epub 2010 Jan 11. PMID 20071021
- [Result] Li HT, Luo S, Trasande L, Hellerstein S, Kang C, Li JX, Zhang Y, Liu JM, Blustein J. Geographic Variations and Temporal Trends in Cesarean Delivery Rates in China, 2008-2014. JAMA. 2017 Jan 3;317(1):69-76. doi: 10.1001/jama.2016.18663. PMID 28030701
- [Result] Zhang Y, Betran AP, Li X, Liu D, Yuan N, Shang L, Lin W, Tu S, Wang L, Wu X, Zhu T, Zhang Y, Lu Z, Zheng L, Gu C, Fang J, Liu Z, Ma L, Cai Z, Yang X, Li H, Zhang H, Zhao X, Yan L, Wang L, Sun X, Luo Q, Liu L, Zhu J, Qin W, Yao Q, Dong S, Yang Y, Cui Z, He Y, Feng X, He L, Zhang H, Zhang L, Wang X, Souza JP, Qi H, Duan T, Zhang J. What is an appropriate caesarean delivery rate for China: a multicentre survey. BJOG. 2022 Jan;129(1):138-147. doi: 10.1111/1471-0528.16951. Epub 2021 Oct 26. PMID 34559941
- [Result] Sharpe EE, Booth JL, Houle TT, Pan PH, Harris LC, Aschenbrenner CA, Eisenach JC. Recovery of physical activity after cesarean delivery and its relationship with pain. Pain. 2019 Oct;160(10):2350-2357. doi: 10.1097/j.pain.0000000000001628. PMID 31145215